CLINICAL TRIAL: NCT06937086
Title: A Phase 3b, Randomized, Multicenter, Controlled Study of Mirikizumab and Placebo or Mirikizumab Concomitantly Administered With Tirzepatide in Adult Participants With Moderately to Severely Active Ulcerative Colitis and Obesity or Overweight
Brief Title: Mirikizumab Administered at the Same Time as Tirzepatide in Adult Participants With Moderately to Severely Active Ulcerative Colitis and Obesity or Overweight: Phase 3b Study
Acronym: COMMIT-UC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27280; 2024-520209-38-00 (EU CTIS Number); I6T-MC-AMCD (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-04-18; First posted 2025-04-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Ulcerative Colitis; Obesity or Overweight
MeSH Terms: conditions — Colitis, Ulcerative; Obesity; Overweight | interventions — mirikizumab; Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Mirikizumab will be open label, tirzepatide and placebo to match will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mirikizumab + Tirzepatide (Experimental): Mirikizumab administered intravenously (IV) then Mirikizumab administered subcutaneously (SC). Tirzepatide administered SC.
  Interventions: Drug: Mirikizumab; Drug: Tirzepatide
- Mirikizumab + Placebo (Experimental): Mirikizumab administered IV then Mirikizumab administered SC. Placebo administered SC.
  Interventions: Drug: Mirikizumab; Drug: Placebo

INTERVENTIONS:
Drug: Mirikizumab — Administered IV
  Other Names: LY3074828
Drug: Mirikizumab — Administered SC
  Other Names: LY3074828
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Mirikizumab + Tirzepatide
Drug: Placebo — Administered SC
  Arms: Mirikizumab + Placebo

SUMMARY:
The main purpose of this study is to show whether in these individuals, treatment with both mirikizumab and tirzepatide, compared with treatment with mirikizumab and placebo, leads to decrease or disappearance of UC symptoms, and loss of at least one-tenth of the overall body weight.

Participation in this study will last up to 61 weeks, including 52 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have had an established diagnosis of UC for ≥3 months before baseline which includes endoscopic evidence of UC and a histopathology report that supports a diagnosis of UC.
* Have moderately to severely active UC as defined by a modified Mayo score (mMS) of 5 to 9 points and endoscopic subscore (ES) of 2 to 3 (confirmed by central review) within 21 days before baseline.
* Participants with a history of UC for greater than or equal to 8 years who have had a surveillance colonoscopy completed within 1 year prior to baseline must have documented negative results for colorectal dysplasia and cancer.
* Have obesity, [body mass index (BMI) 30 kilograms per meter squared (kg/m2)]
* Have overweight (BMI ≥27 kg/m2 to <30 kg/m2) and in the presence of at least 1 of these weight-related comorbid conditions:

  * hypertension
  * Type 2 Diabetes Mellitus (T2DM)
  * dyslipidemia
  * obstructive sleep apnea, or
  * cardiovascular disease.
* Have an inadequate response to, loss of response to, or intolerance to at least 1 of the conventional medication: oral corticosteroids, oral azathioprine (AZA) or 6-mercaptopurine (6-MP), or oral 5-aminosalicylates (for example, mesalamine, sulfasalazine, olsalazine, and balsalazide) and/or who have an inadequate response to or a loss of response to, or are intolerant to advanced therapy for UC, defined as: a biologic or biosimilar medication such as anti-tumor necrosis factor (TNF) antibodies; anti-integrin antibodies, Janus kinase (JAK) inhibitors such as tofacitinib or upadacitinib, sphingosine 1-phosphate receptor 1inhibitors such as etrasimod or ozanimod, or anti-interleukin(IL)-12p40 antibodies, for example, ustekinumab.

Exclusion Criteria:

* Have a current diagnosis of:

  * Crohn's disease
  * inflammatory bowel disease (IBD) unclassified (formerly known as indeterminate colitis), or
  * primary sclerosing cholangitis.
* Have had or will need bowel resection or intestinal or intra-abdominal surgery.
* Have evidence of toxic megacolon, or stricture or stenosis within the colon that cannot be traversed by a sigmoidoscope or colonoscope.
* Have a diagnosis of Type 1 Diabetes Mellitus (T1DM) or have insulin-treated T2DM.
* Have a history of severe hypoglycemia and/or hypoglycemia unawareness within the 6 months prior to screening.
* Have a self-reported change in body weight greater than 5% (gain or reduction) within 3 months prior to screening.
* Have a current or recent acute, active infection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Simultaneously Achieve Clinical Remission and at Least 10% Weight Reduction | Week 52
  Percentage of participants who simultaneously achieve clinical remission and at least 10% weight reduction.

SECONDARY OUTCOMES:
Percentage of Participants Who Achieve Clinical Remission | Week 24 and Week 52
  Percentage of participants who achieve clinical remission.
Percentage of Participants Who Achieve Endoscopic Response | Week 24 and Week 52
  Percentage of participants who achieve endoscopic response.
Percentage of Participants Who Achieve Histologic-Endoscopic Mucosal Improvement Plus Absence of Neutrophils | Week 24 and Week 52
  Percentage of participants who achieve histologic-endoscopic mucosal improvement plus absence of neutrophils
Percentage of Participants Who Achieve Clinical Response | Week 24 and Week 52
  Percentage of participants who achieve clinical response.
Percentage of Participants Who Achieve Endoscopic Remission | Week 24 and Week 52
  Percentage of participants who achieve endoscopic remission.
Percentage of Participants Who Achieve Bowel Movement Urgency Improvement Captured with Urgency Numeric Rating Scale (NRS) | Week 24 and Week 52
  The Urgency NRS is a patient-reported, single-item instrument that measures the severity for the urgency, sudden, or immediate need, to have a bowel movement in the past 24 hours using an 11 point NRS ranging from 0 "no urgency" to 10 "worst possible urgency"
Percentage of Participants Achieving Histologic Remission | Week 24 and Week 52
  Percentage of participants achieving histologic remission.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (191):
- United States (37):
  - Digestive Health Specialists, Dothan, Alabama
  - Smart Cures Clinical Research, Anaheim, California
  - Cedars-Sinai Medical Center, Beverly Hills, California
  - United Medical Doctors - Los Alamitos, Los Alamitos, California
  - California Medical Research Associates, Northridge, California
  - Research Associates of South Florida - Miami - Southwest 8th Street, Miami, Florida
  - Gastro Health Research - Miami, Miami, Florida
  - Orlando Health, Orlando, Florida
  - Digestive and Liver Center of Florida, Orlando, Florida
  - Gastro Health Research - Pensacola, Pensacola, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Grand Teton Research Group, Idaho Falls, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Gastroenterology Health Partners, New Albany, Indiana
  - Gastroenterology Health Partners, Louisville, Kentucky
  - Care Access - New Iberia, New Iberia, Louisiana
  - Louisiana Research Center, Shreveport, Louisiana
  - Capital Digestive Care - Chevy Chase, Chevy Chase, Maryland
  - Lucida Clinical Trials, New Bedford, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - New York Gastroenterology Associates, New York, New York
  - Care Access - Yonkers, Yonkers, New York
  - Coastal Research Institute - Fayetteville, Fayetteville, North Carolina
  - Gastro Intestinal Research Institute of Northern Ohio, LLC, Westlake, Ohio
  - Thomas Jefferson University - Medicine/GI and Hepatology, Philadelphia, Pennsylvania
  - University Gastroenterology - Providence - West River Street, Providence, Rhode Island
  - Gastroenterology Associates - Patewood, Greenville, South Carolina
  - Gastroenterology Center Of The Midsouth, Cordova, Tennessee
  - Gastroenterology Research of San Antonio, San Antonio, Texas
  - Southern Star Research Institute, San Antonio, Texas
  - Tyler Research Institute, Tyler, Texas
  - Gastroenterology Consultants of Southwest Virginia, Roanoke, Virginia
  - Washington Gastroenterology - Tacoma, Tacoma, Washington
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
- Austria (3):
  - Medizinische Universität Graz, Graz
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Medizinische Universität Wien, Vienna
- Belgium (6):
  - AZORG Campus Aalst-Moorselbaan, Aalst
  - Université Libre de Bruxelles - Hôpital Erasme, Brussels
  - AZ Groeninge Campus Kennedylaan, Kortrijk
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège - Domaine Universitaire du Sart Tilman, Liège
  - Clinical Chc Montlégia, Liège
- Brazil (15):
  - NewData Clinical Research - Aracaju, Aracaju
  - L2IP - Instituto de Pesquisas Clínicas, Brasília
  - Loema Instituto de Pesquisa Clinica, Campinas
  - Fundação Universidade de Caxias do Sul (FUCS), Caxias do Sul
  - Centro Digestivo de Curitiba, Curitiba
  - Galileo Medical Research, Juiz de Fora
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - Hospital de Clínicas de Ribeirão Preto, Ribeirão Preto
  - CLIAGEN Clínica de Atenção em Gastroenterologia, Especialidades e Nutrição, Salvador
  - Pesquisare Saude, Santo André
  - CPQuali Pesquisa Clínica, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
  - Clínica Hepatogastro JK, São Paulo
  - CEDOES, Vitória
  - Integral Pesquisa e Ensino, Votuporanga
- Bulgaria (3):
  - University Hospital "St. Ivan Rilski", Gorna Oryahovitsa
  - Multiprofile Hospital for Active Treatment "Knyaginya Klementina" - Sofia EAD, Sofia
  - Medical Center Convex, Sofia
- Canada (5):
  - Victoria Hospital & Children's Hospital - London Health Sciences Centre, London
  - London Digestive Disease Institute, London
  - Clinique IMD, Montreal
  - Vancouver General Hospital, Vancouver
  - (G.I.R.I.) GI Research Institute Foundation, Vancouver
- Czechia (6):
  - SurGal Clinic, Brno
  - Gastroenterologie, Hradec Králové
  - EndoArt, Ostrava
  - ResTrial GastroEndo s.r.o, Prague
  - ISCARE klinické centrum, Prague
  - Masarykova Nemocnice V Usti Nad Labem, Ústí nad Labem
- Denmark (6):
  - Aalborg Universitetshospital, Syd, Aalborg
  - Aarhus Universitetshospital, Skejby, Aarhus
  - Rigshospitalet, Copenhagen
  - Herlev and Gentofte Hospital, Copenhagen
  - Odense Universitetshospital, Odense
  - Vejle Sygehus, Vejle
- France (10):
  - Clinique des Cèdres, Échirolles
  - CHD Vendee, La Roche-sur-Yon
  - Hôpitaux Universitaires Paris Sud - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Chu Saint Eloi, Montpellier
  - Centres Médico Chirurgicaux - Clinique Ambroise Paré, Neuilly-sur-Seine
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet, Nice
  - Hôpital Saint Antoine, Paris
  - Centre Hospitalier Universitaire de Saint Étienne - Hôpital Nord, Saint-Priest-en-Jarez
  - CHU Rangueil, Toulouse
  - Clinique Pasteur, Toulouse
- Germany (6):
  - Universitätsklinikum Frankfurt Goethe-Universität, Frankfurt
  - Praxiszentrum für Gastroenterologie, Grevenbroich
  - Studiengesellschaft BSF Unternehmergesellschaft, Halle
  - Medizinische Hochschule Hannover, Hanover
  - Eugastro GmbH, Leipzig
  - Klinikum Ernst von Bergmann, Potsdam
- Greece (5):
  - Evangelismos General Hospital of Athens, Athens
  - Thoracic General Hospital of Athens "I Sotiria", Athens
  - University General Hospital of Heraklion, Heraklion
  - University Hospital of Ioannina, Ioannina
  - Ippokrateio General Hospital of Thessaloniki, Thessaloniki
- Hungary (3):
  - Semmelweis Egyetem, Budapest
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged
  - CLINFAN Szolgáltató Kft, Szekszárd
- Israel (8):
  - Assuta Ashdod Medical Center, Ashdod
  - Rambam Health Care Campus, Haifa
  - Edith Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
  - Yitzhak Shamir Medical Center, Ẕerifin
- Italy (10):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna
  - Ospedale Specializzato in Gastroenterologia "Saverio de Bellis", Castellana Grotte
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele, Milan
  - Azienda Ospedale - Università Padova, Padua
  - Az. Osp. Ospedali Riuniti VILLA SOFIA-CERVELLO, Palermo
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Ospedale Di Circolo, Rho
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Humanitas, Rozzano
- Mexico (16):
  - San Peregrino Unidad de Investigación, Aguascalientes
  - Scientia Investigacion Clinica S.C., Chihuahua City
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, S.C., Ciudad Madero
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Boca Clinical Trials Mexico S.C., Guadajalara
  - Centro de Investigación Clínica y Medicina Traslacional (CIMeT), Guadalajara
  - Hospital General de Occidente, Guadalajara
  - Health Pharma Querétaro, Juriquilla
  - Centro de Investigación Clinica Chapultepec, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
  - Medical Care and Research SA de CV, Mérida
  - Servicios de Oncología Médica Integral - Monterrey, Monterrey
  - Centro de Investigacion Clinica Chapultepec, Morelia
  - Boca Clinical Trials Mexico SC, Puebla City
  - Clinical Research Institute S.C., Tlalnepantla
  - FAICIC S. de R.L. de C.V., Veracruz
- Netherlands (5):
  - Amsterdam UMC, locatie VUmc, Amsterdam
  - Radboudumc, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (12):
  - Gyncentrum sp. z o.o. NZOZ Holsamed - oddział Libero, Katowice
  - Twoja Przychodnia Opolskie Centrum Medyczne, Opole
  - IRMED, Piotrkow Trybunalski
  - Twoja Przychodnia PCM, Poznan
  - Uniwersyteckie Centrum Stomatologii i Medycyny Specjalistycznej, Poznan
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów
  - Twoja Przychodnia SCM, Szczecin
  - NZOZ GynCentrum - Oddział Warszawa, Warsaw
  - Vivamed Sp. z o.o., Warsaw
  - Medical Network Spółka z o.o. WIP Warsaw IBD Point Profesor Kierkuś, Warsaw
  - Melita Medical, Wroclaw
  - ETG Zamość, Zamość
- CMRC Headlands, LLC, San Juan, Puerto Rico
- Romania (6):
  - Spitalul Județean de Urgență Bacău, Bacau
  - Spitalul Clinic Colentina, Bucharest
  - Spitalul Universitar de Urgență București, Bucharest
  - Constanta County Emergency Clinical Hospital Sf.Ap.Andrei, Constanța
  - Spitalul Clinic Județean de Urgență, Craiova
  - S.C Centrul de Gastroenterologie Dr. Goldis S.R.L, Timișoara
- Zemun Medical Centre, Zemun, Serbia
- Slovakia (4):
  - Fakultna nemocnica s poliklinikou F.D.Roosevelta Banska Bystrica, Banská Bystrica
  - Cliniq s.r.o., Bratislava
  - ENDOMED, Košice
  - Gastro LM, Prešov
- Spain (10):
  - Centro Médico Teknon, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Complejo Hospitalario Universitario de Ferrol (CHUF)- Hospital Arquitecto Marcide, Ferrol
  - Hospital de Cabueñes, Gijón
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Turkey (Türkiye) (9):
  - Gazi University Health Research and Application Center Gazi Hospital, Ankara
  - Antalya Egitim ve Arastırma Hastanesi, Antalya
  - Uludag Universitesi, Bursa
  - Eskisehir Osmangazi University, Eskişehir
  - Mustafa Kemal Universitesi, Hatay
  - Bezmialem Vakf Üniversitesi, Istanbul
  - Ege Universitesi Hastanesi, Izmir
  - Kocaeli University Medical Faculty Hospital, İzmit
  - Mersin University, Mersin
- United Kingdom (4):
  - Southmead Hospital, Bristol
  - Ninewells Hospital and Medical School, Dundee
  - Royal Devon & Exeter Hospital, Exeter
  - Royal London Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal should be approved by an independent review panel and researchers should sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: Related Info — https://trials.lilly.com/en-US/trial/600155